CLINICAL TRIAL: NCT07122713
Title: Multi-institutional Prospective Pilot Study of Definitive Breast Radiation Therapy for Invasive Breast Cancer Patients Not Undergoing Definitive Surgery
Brief Title: Definitive Radiation Therapy for Inoperable Breast Cancer
Acronym: DEFINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexander Stessin (Other)
Collaborators: Northwell Health (Other)
Responsible Party: Sponsor-Investigator, Alexander Stessin, Professor, Department of Radiation Oncology, Stony Brook University
Organization: Stony Brook University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBU-BREAST-DEFINE; IRB2024-00364 (Other: Stony Brook University)
Record Dates: First submitted 2025-07-24; First posted 2025-08-14 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Breast Adenocarcinoma
Keywords: inoperable breast cancer; radiation therapy; breast radiation; novel treatment; new treatment breast; cyberknife; non-invasive; stereotactic radiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- A: Ipsilateral axillary node-negative breast cancer (Experimental): Patients with ipsilateral axillary lymph node-negative disease, regardless of metastatic status (Stages T1-4 N0 M0-1)
  Interventions: Radiation: Whole breast radiation with simultaneous integrated boost (WB-SIB) to primary breast tumor
- B: Ipsilateral axillary node-positive breast cancer (Experimental): Patients with ipsilateral axillary node-positive disease, regardless of metastatic status (Stages T1-4 N1-2 M0-1)
  Interventions: Radiation: Whole breast radiation with simultaneous integrated boost (WB-SIB) to primary breast tumor and ipsilateral axillary lymph nodes

INTERVENTIONS:
Radiation: Whole breast radiation with simultaneous integrated boost (WB-SIB) to primary breast tumor — Radiation with 26Gy to the whole breast and 40Gy simultaneous integrated boost to gross disease in the breast, in five fractions
  Arms: A: Ipsilateral axillary node-negative breast cancer
Radiation: Whole breast radiation with simultaneous integrated boost (WB-SIB) to primary breast tumor and ipsilateral axillary lymph nodes — Radiation with 26Gy to the whole breast and regional nodes with a 40Gy simultaneous integrated boost to gross disease in breast and ipsilateral axillary nodal areas, in five fractions
  Arms: B: Ipsilateral axillary node-positive breast cancer

SUMMARY:
The purpose of this study is to find out if adding radiation therapy to routine medications for breast cancer helps in reducing and preventing the cancer from getting worse. Patients with a locally advanced breast cancer who cannot, or do not want to, undergo surgery are eligible to participate. Participation in this study does not prevent you from undergoing surgery in the future.

DETAILED DESCRIPTION:
Patients who cannot undergo surgical resection for either breast cancer or local control of metastatic cancer have limited effective treatment options. Treatments typically employed in the adjuvant setting have been found in the definitive setting to be inferior to surgery followed by adjuvant therapy. This raises the necessity of evaluating the use of ablative doses of radiation to provide durable local control of the tumor in such patients. Indeed, there is growing evidence that RT is effective in the adjuvant setting. This is a study of concurrent ultra-hypofractionated whole breast whole breast radiation delivered via simultaneous integrated boost to the gross tumor for breast cancer patients not undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven invasive carcinoma of the breast, either lobular, ductal and/or no special type
* T1-T4, N0-2, M0-1 invasive breast carcinoma by radiological or clinical criteria
* Cancer is deemed unresectable, or the patient is a poor surgical candidate as determined following evaluation by a surgeon, or patient declines surgery.
* Life expectancy > 6 months
* Negative pregnancy test at the time of start of treatment in any female of reproductive age

Exclusion Criteria:

* Concurrent systemic therapy (except for endocrine therapy, HER2-targeted therapy, or immunotherapy which are permitted)
* Prior radiation to ipsilateral breast or regional nodes
* Inability to receive study treatment planning and treatment secondary to body habitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2033-12-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Safety | 12 months
  Incidence of physician-assessed treatment-related toxicity ≥ Grade 4 events, as defined using CTCAE 5.0

SECONDARY OUTCOMES:
Acute Toxicity | 12 months
  Percent of participants with any physician-assessed treatment-related Grade 1-5 events using CTCAE 5.0. Grade 1 events are limited to fatigue, skin, breast, ribs, heart and lungs.
Late Toxicity | 5 years
  Percent of participants with any physician-assessed treatment-related Grade 2-5 events using CTCAE 5.0.
Treatment Tolerability by EORTC QLQ-C30 | 2 years
  Patient reported quality of life measured using the quality of life questionnaire C30 (QLQ-C30), developed by the European Organisation for Research and Treatment of Cancer. This scale includes 5 functional and 3 symptom scales, each scored as a 0-100 scale, where higher scores indicate a better outcome on functional scales and global health status, and a worse outcome on symptoms.
Treatment Tolerability by EORTC QLQ-BR42 | 2 years
  Patient reported quality of life measured using the quality of life questionnaire BR42 (QLQ-BR42), developed by the European Organisation for Research and Treatment of Cancer. This scale assesses symptoms, body image and sexual functioning scales, each scored as a 0-100 scale, where higher scores indicate worse outcome on symptoms.
Tumor Response Rate in the Gross Disease Volume (40Gy) | 1 year
  Measured on follow-up MRI or CT imaging using RECIST criteria
Progression Free Rate in the Microscopic Disease Volume (26Gy) | 1 year
  Measured on follow-up MRI or CT imaging using RECIST criteria
Clinical Response in patients with Palpable Disease | 1 year
  Caliper measurements (2-dimensional)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stessin, MD PhD, Principal Investigator — Stony Brook University Hospital
Locations (1):
- Stony Brook University Cancer Center, Stony Brook, New York, United States